CLINICAL TRIAL: NCT04177342
Title: Influence of Intraoperative Opioids (Oxycodone/Fentanyl) Usage on the Post-operative Pain Management of Peroral Endoscopic Myotomy (POEM)
Brief Title: Post Operative Pain Control of POEM Procedure
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chen Wannan (Other)
Responsible Party: Sponsor-Investigator, Chen Wannan, Principal Investigator, Shanghai Zhongshan Hospital
Organization: Shanghai Zhongshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: POEM pain control
Record Dates: First submitted 2019-04-02; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Achalasia
Keywords: achalasia; Peroral endoscopic myotomy; post-operative pain
MeSH Terms: conditions — Esophageal Achalasia; Pain, Postoperative | interventions — Fentanyl; Oxycodone

STUDY DESIGN:
Intervention Model Description: patients will be devided randomly into two groups. One group will be given oxycodone and the other will be given fentanyl during the POEM procedure. Post procedure pain condition will be recorded.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- fentanyl (Active Comparator): the patients use remifentanil and fentanyl as intra-operatively pain control and compare the post-operative pain condition with the oxycodone group
  Interventions: Drug: Fentanyl
- oxycodone (Experimental): the patients use oxycodone and remifentanil as intra-operatively pain control and compare the post-operative pain condition with the fentanyl group
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Fentanyl — the patients use remifentanil and fentanyl as intra-operatively pain control and compare the post-operative pain condition with the oxycodone group
  Arms: fentanyl
Drug: Oxycodone — the patients use oxycodone and remifentanil as intra-operatively pain control and compare the post-operative pain condition with the fentanyl group
  Arms: oxycodone

SUMMARY:
Peroral endoscopic myotomy (POEM) is a minimally invasive treatment for esophageal achalasia with a natural orifice transluminal endoscopic procedure and far less invasive than the standard surgical or laparoscopic Heller myotomy (LHM). Less is known about the postoperative pain after POEM and the minor surgery trauma, short length of stay may lead to underestimation of postoperative pain control. We tend to observe the pain status after the POEM surgery under the empirical treatment in our center, and find a proper intra-operative way of pain control to solve the post-operative pain and seek the possible influence factors of postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Achalasia patients undergoing elective POEM surgery
* age 18-80
* BMI 18-30 kg/m2

Exclusion Criteria:

* Patient refusal
* ASA≥ 3
* abnormality of liver and kidney function in patients
* patients with mental disorder, language disorder, and other patients who can not cooperate with and complete the follow-up and questionnaire pre- and post- operatively
* patients (including propanotamo, propofol, lidocaine, and other drugs) against drug taboos in the anesthetic scheme
* patients with chronic pain before operation with analgesic drugs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
post-operative pain condition | 36 hours after the POEM surgery
  use Visual Analogue Scale/Score(0-10) to record post operative pain
post-operative PCA usage volumn | 36 hours after the POEM surgery
  record PCA usage volumn(ml) to see the dosage of opiods used after the surgery
post-operative sleep quality | 48 hoursafter the surgery
  Postoperative sleep quality was investigated with a self-reported sleep questionnaire including 6 yes/no questions(0-6) with full score 6 represented the worst sleep

SECONDARY OUTCOMES:
chronic pain condition | 28 days after discharge
  use Visual Analogue Scale/Score(0-10) to evaluate the pain condition

CONTACTS AND LOCATIONS:
Overall Officials: Wannan Chen, MD, Principal Investigator — Shanhai Zhongshan